CLINICAL TRIAL: NCT02770222
Title: A Single-center, Open-label, Randomized, Two-part, Two-treatment, Two-period Crossover Study to Investigate the Effect of Gemfibrozil or Rifampicin on the Pharmacokinetics of Selexipag and Its Metabolite ACT-333679 in Healthy Male Subjects.
Brief Title: A Clinical Study to Investigate the Effect of Gemfibrozil or Rifampicin on Blood Concentrations of Selexipag in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-065-113; 2016-000811-34 (EudraCT Number)
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics
MeSH Terms: interventions — selexipag; Gemfibrozil; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1, sequence AB (Experimental): Subjects participate in two study periods: During the first period (Treatment A), they receive oral selexipag on Day 1. During the second period (Treatment B), they receive multiple oral dose of gemfibrozil from Day 1 to Day 9. Subjects also receive a single oral dose of selexipag on Day 4 concomitantly with gemfibrozil. There is a washout period of 14 to 21 days between the two periods.
  Interventions: Drug: Selexipag; Drug: Gemfibrozil
- Part 1, sequence BA (Experimental): Subjects participate in two study periods: During the first period (Treatment B), they receive multiple oral dose of gemfibrozil from Day 1 to Day 9. They also receive a single oral dose of selexipag on Day 4 concomitantly with gemfibrozil. During the second period (Treatment A) they receive oral selexipag on Day 1. There is a washout period of 14 to 21 days between the two periods.
  Interventions: Drug: Selexipag; Drug: Gemfibrozil
- Part 2, sequence AB (Experimental): Subjects participate in two study periods: During the first period (Treatment A), they receive oral selexipag on Day 1. During the second period (Treatment B), they receive rifampicin once daily from Day 1 to Day 9. Subjects also receive a single oral dose of selexipag on Day 7 together with the dose of rifampicin.There is a washout period of 14 to 21 days between the two periods.
  Interventions: Drug: Selexipag; Drug: Rifampicin
- Part 2, sequence BA (Experimental): Subjects participate in two study periods: During the first period (Treatment B), they receive rifampicin once daily from Day 1 to Day 9. Subjects also receive a single oral dose of selexipag on Day 7 together with the dose of rifampicin. During the second period (Treatment A), they receive oral selexipag on Day 1. There is a washout period of 14 to 21 days between the two periods.
  Interventions: Drug: Selexipag; Drug: Rifampicin

INTERVENTIONS:
Drug: Selexipag — Two selexipag film-coated tablets of 200 µg as single oral dose (total dose = 400 µg)
  Other Names: ACT-293987
Drug: Gemfibrozil — Gemfibrozil film-coated tablet of 600 mg administered orally b.i.d. from Day 1 to Day 9
  Arms: Part 1, sequence AB; Part 1, sequence BA
Drug: Rifampicin — Rifampicin film-coated tablet of 600 mg administered orally o.d.from Day 1 to Day 9
  Arms: Part 2, sequence AB; Part 2, sequence BA

SUMMARY:
The primary objectives of this 2-part drug interaction study are as follows:

* To evaluate the effect of gemfibrozil on the pharmacokinetics (i.e., amount in the blood) of selexipag and its metabolite ACT-333679 (Part I).
* To evaluate the effect of rifampicin on the pharmacokinetics of selexipag and its metabolite ACT-333679 (Part II).

DETAILED DESCRIPTION:
Because non-clinical studies have shown that selexipag and its active metabolite, ACT-333679, are substrates for cytochrome P450 2C8 (CYP2C8), the present clinical study aims at investigating the effect of a strong inhibitor (gemfibrozil) and a moderate inducer (rifampicin) of CYP2C8 on the pharmacokinetic of selexipag and ACT-333679 as recommended by the FDA's Guidance for Industry Drug Interaction Studies (FDA, 2012).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male subjects aged between 18 and 55 years (inclusive) at screening.
* Body mass index of 18.0 to 28.0 kg/m2 (inclusive) at screening.
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests at screening.

Exclusion Criteria:

* Any contraindication to gemfibrozil or rifampicin treatment.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might put the subject at risk of participation in the study or interfere with the absorption, distribution, metabolism or excretion of the study treatments.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to infinity [AUC(0-inf)] of selexipag and ACT-333679 | Blood samples at different time points from pre-dose up to 72 hours after selexipag administration in each study period (except for the period with co-administration of gemfibrozil: up to 144 hours)
  AUC(0-inf) is calculated for selexipag and its metabolite, ACT-333679, following administration of selexipag alone or concomitantly with gemfibrozil (Part I) or rifampicin (Part II)
Maximum plasma concentration (Cmax) of selexipag and ACT-333679 | Blood samples at different time points from pre-dose up to 72 hours after selexipag administration in each study period (except for the period with co-administration of gemfibrozil: up to 144 hours)
  Cmax is directly derived from the individual plasma concentration-time curves for selexipag and its metabolite, ACT-333679, following administration of selexipag alone or concomitantly with gemfibrozil (Part I) or rifampicin (Part II)

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification [(AUC(0-t)] of selexipag and ACT-333679 | Blood samples at different time points from pre-dose up to 72 hours after selexipag administration in each study period (except for the period with co-administration of gemfibrozil: up to 144 hours)
  AUC(0-t) is calculated for selexipag and ACT-333679,following administration of selexipag alone or concomitantly with gemfibrozil (Part I) or rifampicin (Part II)
Time to reach maximum plasma concentration (tmax) of selexipag and ACT-333679 | Blood samples at different time points from pre-dose up to 72 hours after selexipag administration in each study period (except for the period with co-administration of gemfibrozil: up to 144 hours)
  tmax is directly derived from the individual plasma concentration-time curves for selexipag and its metabolite, ACT-333679, following administration of selexipag alone or concomitantly with gemfibrozil (Part I) or rifampicin (Part II)
Terminal elimination half-life (t1/2) of selexipag and ACT-333679 | Blood samples at different time points from pre-dose up to 72 hours after selexipag administration in each study period (except for the period with co-administration of gemfibrozil: up to 144 hours)
  t1/2 is the period of time required for the concentration levels of selexipag or ACT-333679 to be reduced by one-half, following administration of selexipag alone or concomitantly with gemfibrozil (Part I) or rifampicin (Part II)

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events and serious adverse events | Up to 35 days (from first study drug administration to end of study visit)
  A treatment-emergent AE is any AE temporally associated with the use of a study treatment, whether or not considered related to the study treatment
Incidence of safety events of interest | Up to 35 days (from first study drug administration to end of study visit)
  Include any abnormalities in ECG, vital signs or laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Bruderer, PhD, Study Director — Actelion

REFERENCES:
- [Derived] Bruderer S, Petersen-Sylla M, Boehler M, Remenova T, Halabi A, Dingemanse J. Effect of gemfibrozil and rifampicin on the pharmacokinetics of selexipag and its active metabolite in healthy subjects. Br J Clin Pharmacol. 2017 Dec;83(12):2778-2788. doi: 10.1111/bcp.13379. Epub 2017 Aug 16. PMID 28715853